CLINICAL TRIAL: NCT03033121
Title: More Favorable Metabolic Impact of Three-times-weekly Versus Daily Growth Hormone (GH) Treatment in naïve GH-deficient Children
Brief Title: Three-times-weekly Versus Daily Growth Hormone (GH) Treatment in naïve GH-deficient Children
Acronym: GH 3 wk dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Carla Giordano, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-wk-GH
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Growth Hormone Treatment
Keywords: growth hormone; children; metabolism
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Active Comparator): Sixteen growth hormone (GH) deficiency children were assigned to receive daily growth hormone therapy for 12 months. The investigators used an initial weekly dose of 0.175 mg/kg (corresponding to the daily dose of 0.025 mg/Kg) of GH with a gradual increase every 6 months in order to always maintain the insulin growth factor (IGF)-I levels in the normal range. In detail, from months 1 to 6 the investigators used the mean weekly dose of 0.175 mg/kg and from months 6 to 12 the mean weekly dose of 0.20 mg/kg.
  Interventions: Drug: Growth Hormone
- group B (Active Comparator): Sixteen growth hormone (GH) deficiency children were assigned to receive three time weekly growth hormone therapy for 12 months. The investigators used an initial weekly dose of 0.175 mg/kg (corresponding to the daily dose of 0.025 mg/Kg) of GH with a gradual increase every 6 months in order to always maintain the insulin growth factor (IGF)-I levels in the normal range. In detail, from months 1 to 6 the investigators used the mean weekly dose of 0.175 mg/kg and from months 6 to 12 the mean weekly dose of 0.20 mg/kg.
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone

SUMMARY:
Growth hormone (GH) treatment in patients with GH deficiency (GHD) is commonly administered daily, although the pulsatile GH secretion is unlikely to be achieved and this regimen is often not complied. The auxological effect of three injections per week (TIW) regimen is controversial, while the metabolic effects were never evaluated in children. The objective of this study was to evaluate whether two different regimens of weekly injections could lead to similar auxological and metabolic effects in children with GHD.

DETAILED DESCRIPTION:
Thirty-two children with growth hormone (GH) deficiency (25 males, mean age 10.5 ± 2.2 yr) were randomly assigned to receive daily (group A, No 16) or three injections per week (group B, No 16) GH therapy for 12 months.

Auxological parameters, insulin-like growth factor-I (IGF-I), glucose and insulin during an oral glucose tolerance test, glycosylated hemoglobin, lipid profile, the oral disposition index (DIo), the homeostasis model assessment estimate of insulin resistance (Homa-IR), the quantitative insulin sensitivity check index (QUICKI) and the insulin sensitivity index (ISI) were evaluated in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone deficiency clinically and biochemically demonstrated

Exclusion Criteria:

* Children affected by multiple pituitary hormone deficiency or receiving any other kind of hormonal replacement therapy or drug and GHD children with a shorter follow-up

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-01-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
height | 12 months
  height (standard deviation)
weight | 12 months
  weight (kilograms)
body mass index | 12 months
  body mass index (kilograms/m2)
Insulin growth factor-I | 12 months
  insulin growth factor (IGF)-I (ug/L)
glucose | 12 months
  glucose (mmol/l) during oral glucose tolerance test
insulin | 12 months
  insulin (uU/ml) during oral glucose tolerance test
glycated hemoglobin | 12 months
  glycated hemoglobin (%)
ISI Matsuda | 12 months
  Insulin Sensitivity Index
Oral disposition index | 12 months
  Oral Disposition Index (DIo)
Homa IR | 12 months
  The homeostatic model assessment of insulin resistance
LDL cholesterol | 12 months
  Low Density Lipoprotein cholesterol (mmol/l)
Triglycerides | 12 months
  triglycerides (mmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology - University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ciresi A, Ciccio F, Radellini S, Guarnotta V, Calcaterra AM, Giordano C. More Favorable Metabolic Impact of Three-Times-Weekly versus Daily Growth Hormone Treatment in Naive GH-Deficient Children. Int J Endocrinol. 2017;2017:8469680. doi: 10.1155/2017/8469680. Epub 2017 May 28. PMID 28634491